CLINICAL TRIAL: NCT07037212
Title: The Impact of Intensive Medical Nutrition Therapy on Glycemic Control, Inflammation, and Gut Barrier Regulation in Adults With Type 2 Diabetes Mellitus: a RCT
Brief Title: Intensive Medical Nutrition Therapy in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serap Balaban Barta (Other)
Responsible Party: Sponsor-Investigator, Serap Balaban Barta, Dr. Researcher, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/095-2020085
Record Dates: First submitted 2025-06-08; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Systemic Inflammation; Intestinal Permeability; Glycemic Control
Keywords: Type 2 Diabetes Mellitus; Medical nutrition therapy; Glycemic control; Inflammation; Zonulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups: an intensive medical nutrition therapy (MNT) group receiving individualized MNT with weekly follow-ups for 12 weeks, and a control group receiving standard dietary advice in a single session. Both groups will be followed concurrently.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive MNT group (Experimental): Participants in this group will receive individualized intensive medical nutrition therapy (MNT) with weekly in-person follow-ups and dietary counseling for 12 weeks. The MNT is tailored based on patient characteristics and focuses on improving glycemic control, reducing inflammation, and enhancing gut barrier function.
  Interventions: Behavioral: Intensive Medical Nutrition Therapy (MNT)
- Control group (Active Comparator): Participants in this group will receive standard dietary advice in a single counseling session at baseline. No further follow-up or dietary intervention will be provided during the study period.
  Interventions: Behavioral: Standard Dietary Counseling

INTERVENTIONS:
Behavioral: Intensive Medical Nutrition Therapy (MNT) — Participants will receive individualized intensive medical nutrition therapy (MNT) with weekly dietary counseling and follow-ups for 12 weeks. The intervention focuses on improving glycemic control, reducing systemic inflammation, and enhancing gut barrier function.
  Arms: Intensive MNT group
Behavioral: Standard Dietary Counseling — Participants will receive standard dietary advice in a single counseling session at baseline. No further dietary intervention will be provided.
  Arms: Control group

SUMMARY:
This study aims to investigate the effects of intensive medical nutrition therapy on blood sugar control, systemic inflammation, and gut barrier function in adults with type 2 diabetes mellitus. In this randomized controlled trial, adults with type 2 diabetes mellitus will be assigned to either an intensive medical nutrition therapy group or a control group. The intensive medical nutrition therapy group will receive individualized nutrition therapy and weekly follow-ups for 12 weeks, while the control group will receive standard dietary counseling. The study will assess changes in glycemic control (HbA1c, fasting plasma glucose), inflammatory markers (TNF-α, IL-6), and intestinal permeability (ZO-1), as well as quality of life and self-care behaviors. The goal is to evaluate whether intensive medical nutrition therapy can improve metabolic outcomes and overall health in adults with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus is associated with systemic inflammation, insulin resistance, and increased intestinal permeability, all of which contribute to disease progression and complications. Intensive medical nutrition therapy has been proposed as a non-pharmacological strategy to improve glycemic control and reduce inflammation. This randomized controlled trial evaluates the impact of a 12-week intensive medical nutrition therapy program on glycemic control, inflammatory markers, and gut barrier function in adults with type 2 diabetes mellitus. Participants will be randomized into two groups: an intensive MNT group receiving individualized dietary counseling with weekly follow-ups, and a control group receiving standard dietary advice. The study will assess changes in fasting plasma glucose, HbA1c, TNF-α, IL-6, and zonulin (ZO-1) levels, along with quality of life and diabetes self-care behaviors. The findings will provide insights into the potential role of medical nutrition therapy in modulating inflammation-related pathways and improving metabolic outcomes in adults with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM) for at least one year
* Age 20 to 65 years
* Body Mass Index (BMI) ≥ 25 kg/m²
* Currently receiving oral anti-diabetic (OAD) medications
* HbA1c ≥ 7%
* Able and willing to provide written informed consent

Exclusion Criteria:

* Receiving insulin therapy
* Presence of uncontrolled comorbid conditions (advanced cardiovascular disease, cerebrovascular disease, severe kidney disease, cancer, or diabetes-related vision impairment)
* Presence of acute infection
* Taking antioxidant vitamins or mineral supplements
* Diagnosed with cognitive impairment or dementia
* Using medical devices such as pacemakers or hearing aids
* Currently participating in another dietary program
* Pregnant or breastfeeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (%) | From enrollment to the end of treatment at 12 weeks
  Change in hemoglobin A1c (%) from baseline to 12 weeks.
Change in Fasting Plasma Glucose | From enrollment to the end of treatment at 12 weeks
  Change in fasting glucose levels (mg/dL) from baseline to 12 weeks.

SECONDARY OUTCOMES:
Change in TNF-α | From enrollment to the end of treatment at 12 weeks
  Change in serum tumor necrosis factor-alpha (TNF-α) levels, measured by ELISA, from baseline to 12 weeks.
Change in IL-6 | From enrollment to the end of treatment at 12 weeks
  Change in serum interleukin-6 (IL-6) levels, measured by ELISA, from baseline to 12 weeks.
Change in Zonulin | From enrollment to the end of treatment at 12 weeks
  Change in serum zonulin (ZO-1) levels, as a marker of intestinal permeability, measured by ELISA, from baseline to 12 weeks.
Change in Body Weight | From enrollment to the end of treatment at 12 weeks
  Change in body weight (in kilograms), measured using a calibrated digital scale. Measurements are taken with participants wearing light clothing and no shoes, under fasting conditions. Body weight will be recorded at baseline and at 12 weeks. Body weight is used as a reference value for BMI.
Change in Height | From enrollment to the end of treatment at 12 weeks
  Change in participant height (in meters), measured using a stadiometer while participants are barefoot and standing upright in the Frankfurt plane. Height will be recorded at baseline and at 12 weeks.
  Height is used as a reference value for BMI.
Change in Body Mass Index (BMI) | From enrollment to the end of treatment at 12 weeks
  Body weight and height were used to calculate BMI (kg/m²). Change in BMI from baseline to 12 weeks will be reported.
Change in Diabetes-related Quality of Life | From enrollment to the end of treatment at 12 weeks
  Change in total score on the Diabetes Quality of Life (DQOL) questionnaire, which ranges from 0 to 135.
  Higher scores indicate better quality of life. The DQOL includes 45 items covering treatment satisfaction (15 items), psychological impact of the treatment (19 items), concerns/anxieties about the future course and effects of the disease (4 items), and social and occupational concerns/anxieties (7 items).
  Scores are calculated at baseline and at 12 weeks.
Change in Self-Care Behaviors | From enrollment to the end of treatment at 12 weeks
  Change in total score on the Summary of Diabetes Self-Care Activities (SDSCA) measure, which ranges from 0 to 7.
  Higher scores indicate a higher frequency of self-care behaviors. The SDSCA consists of four subscales- diet (4 items), exercise (2 items), blood glucose monitoring (2 items), and foot care (2 items) with a total of 10 questions.
Change in Physical Activity Score | From enrollment to the end of treatment at 12 weeks
  Change in total physical activity level, assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF).
  The score is calculated in MET-minutes/week based on participant-reported duration and frequency of walking, moderate, and vigorous physical activities over the past 7 days.
  Scores typically range from 0 to over 10,000 MET-min/week. Higher scores indicate greater levels of physical activity.
  Categories:
  Inactive (<600 MET-min/week)
  Minimally Active (600-3000 MET-min/week)
  Active (>3000 MET-min/week)

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Medical Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No